CLINICAL TRIAL: NCT07019831
Title: Imaging the Respiratory Effects of Truncal Adiposity in Healthy Subjects
Brief Title: A Study of Body Fat Distribution and Airway Mechanics in Healthy Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maurizio F. Cereda, MD (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor-Investigator, Maurizio F. Cereda, MD, Associate Professor of Anesthesia, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025P001553
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers Only
Keywords: obesity; electrical impedance tomography; computed tomography; esophageal manometry; airway geometry
MeSH Terms: conditions — Obesity | interventions — Posture; Supine Position; Prone Position

STUDY DESIGN:
Intervention Model Description: In a prospective, single-center, physiological, crossover study, the investigators will recruit 20 healthy volunteers across four standard body mass index categories (normal weight, overweight, class I obesity, class II/III obesity).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, respiratory mechanics and adipose distribution in two body positions (Experimental): A total of 20 healthy volunteers will undergo assessments of respiratory mechanics in the supine and prone position. Then, the same subjects will undergo CT scans of the lungs in both positions. Body positions will be randomly applied for 15 minutes each.
  Interventions: Procedure: Body positioning

INTERVENTIONS:
Procedure: Body positioning — Each subject will breathe in both the supine and prone positions, randomly applied for 15 minutes each. The procedure will be performed twice: once for the assessment of respiratory physiology, and once for computed tomography acquisition.
  Other Names: Supine and prone

SUMMARY:
This study investigates how body fat distribution affects airway closure and lung mechanics in healthy adults. Using Electrical Impedance Tomography (EIT), esophageal manometry, and computed tomography (CT), we aim to characterize how varying BMI and fat topography influence regional ventilation and airway collapse in supine and prone positions. Healthy volunteers with a range of BMIs will undergo a 2-hour imaging session with noninvasive and minimally invasive monitoring.

DETAILED DESCRIPTION:
This physiological research study explores the relationship between body habitus, fat distribution, and mechanical responses of the lung to the prone and supine position. In a prospective, single-center, physiological, crossover study, study subjects (n=20) will be recruited among healthy volunteers across BMI categories. Lung function will be assessed in the supine and prone position (maintained for 15 min). Intrathoracic pressure (ITP) will be measured using esophageal manometry. Airway opening pressure (AOP) will be measured by as the airway pressure (non-invasively applied through a mask) needed to match ITP. Regional ventilation will be measured in both positions using electrical impedance tomography. Subjects will then transfer to the computed tomography (CT) scanner, where supine and prone images will be acquired during breath holds after normal expiration and after full inspiration. CT scans will then be analyzed for the quantification of lung volumes, thoracic adipose mass and airway geometry.

ELIGIBILITY:
Inclusion Criteria

• Healthy subjects older than 18 years and younger than 80.

Exclusion Criteria

* Pre-existing cardiopulmonary disease
* history of tobacco or ecigarette smoking

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2028-01-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Lung volumes | Day 1, 15 minutes after breathing in the supine and in the prone position
  Lung volumes will be measured from quantitative analysis of CT scans obtained in the supine and in the prone position.

SECONDARY OUTCOMES:
Thoracic adiposity | Day 1
  Thoracic adipose tissue will be quantified from analysis of computed tomography images as area of adipose tissue (cm^2) at multiple vertebral levels.

OTHER OUTCOMES:
Airway diameters | Day 1, after 15 minutes in the supine and prone positions
  CT scans will be digitally processed for the identification of airway branches down to the 4th bronchial generation. Bronchial cross sectional areas will then be measured (mm^2) and compared between body positions.
Intrathoracic pressure (ITP) | Day 1, after 15 minutes in the supine and prone positions.
  ITP (cmH2O) will be measured as the pressure in the esophagus at the end of expiration. This will be obtained through a thin balloon mounted catheter placed in the distal esophagus through a nostril.
Airway opening pressure (AOP) | Day 1, after 15 minutes in supine and prone position
  AOP (cmH2O) will be measured as the airway pressure that matches ITP during the graded application of positive airway pressure through a face mask.
Regional ventilation | Day 1, after 15 minutes in the supine or prone position
  Changes in EIT-derived measurements of regional ventilation with PEEP titration and prone positioning. EIT regional ventilation is measured as percentage of total ventilation in each examined lung region.
Age | Day 1
  Age will be measured in years and obtained during subject interview
Height | Day 1
  Body height will be measured in meters and will be aggregated with body weight to yield body mass index (BMI) in kg/m^2.
Weight | Day 1
  Body weight will be measured in kg and will be aggregated with height to yield body mass index (BMI) in kg/m^2
Thoracic circumference | Day 1
  Thoracic circumference will be measured in cm using a tape ruler placed at nipple level.
Abdominal circumference | Day 1
  Abdominal circumference will be measured in cm using a tape ruler at the level of the umbilicus.
Hip circumference | Day 1
  Hip circumference will be measured in cm using a tape ruler placed around the widest portion of the hips.
Medical history | Day 1
  During subject interview, the presence of the following conditions will be recorded: hypertension, diabetes, asthma.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spina S, Mantz L, Xin Y, Moscho DC, Ribeiro De Santis Santiago R, Grassi L, Nova A, Gerard SE, Bittner EA, Fintelmann FJ, Berra L, Cereda M. The pleural gradient does not reflect the superimposed pressure in patients with class III obesity. Crit Care. 2024 Sep 16;28(1):306. doi: 10.1186/s13054-024-05097-6. PMID 39285477
- [Background] Giani M, Restivo A, Raimondi Cominesi D, Fracchia R, Pozzi M, Del Sorbo L, Foti G, Brochard L, Rezoagli E. Prone-position decreases airway closure in a patient with ARDS undergoing venovenous extracorporeal membrane oxygenation. J Clin Monit Comput. 2024 Dec;38(6):1425-1429. doi: 10.1007/s10877-024-01182-x. Epub 2024 Jul 27. PMID 39066871
- [Background] Coudroy R, Vimpere D, Aissaoui N, Younan R, Bailleul C, Couteau-Chardon A, Lancelot A, Guerot E, Chen L, Brochard L, Diehl JL. Prevalence of Complete Airway Closure According to Body Mass Index in Acute Respiratory Distress Syndrome. Anesthesiology. 2020 Oct 1;133(4):867-878. doi: 10.1097/ALN.0000000000003444. PMID 32701573
- [Background] Jones RL, Nzekwu MM. The effects of body mass index on lung volumes. Chest. 2006 Sep;130(3):827-33. doi: 10.1378/chest.130.3.827. PMID 16963682
- [Background] Florio G, De Santis Santiago RR, Fumagalli J, Imber DA, Marrazzo F, Sonny A, Bagchi A, Fitch AK, Anekwe CV, Amato MBP, Arora P, Kacmarek RM, Berra L. Pleural Pressure Targeted Positive Airway Pressure Improves Cardiopulmonary Function in Spontaneously Breathing Patients With Obesity. Chest. 2021 Jun;159(6):2373-2383. doi: 10.1016/j.chest.2021.01.055. Epub 2021 May 8. PMID 34099131